CLINICAL TRIAL: NCT04627012
Title: The Effectiveness and Safety of Lenvatinib Combined Anti-programmed Death Immunotherapy for the Advanced Hepatocellular Carcinoma
Brief Title: Lenvatinib Combined Anti-PD1 Antibody for the Advanced Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, MD, Sun Yat-sen University
Other Study IDs: GYEYJR-2
Record Dates: First submitted 2020-11-08; First posted 2020-11-13 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma; Anti-PD1 Antibody; Liver Diseases
Keywords: Tislelizumab; Lenvatinib; Toripalimab; Sintilimab; Camrelizumab; Keytruda; Opdivo
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Diseases | interventions — lenvatinib; Nivolumab; camrelizumab; pembrolizumab; toripalimab; sintilimab; tislelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Lenvatinib — 12 mg (or 8 mg) once daily (QD) oral dosing.
Drug: Opdivo — 3mg/mg intravenously every 3 weeks
Drug: Camrelizumab — 200mg intravenously every 3 weeks
Drug: Keytruda — 200mg intravenously every 3 weeks
Drug: Toripalimab — 240mg intravenously every 3 weeks
Drug: Sintilimab — 200mg intravenously every 3 weeks
Drug: Tislelizumab — 200mg intravenously every 3 weeks

SUMMARY:
For the advanced hepatocellular carcinoma (HCC), the targeted therapy and immunotherapy are recommended. This study focused on the management of Lenvatinib combined anti-PD1 antibody for the HCC. This study will create a database that will provide clinical parameters and outcomes of patients undergoing Lenvatinib and anti-PD1 antibody as part of their standard of care in hopes of answering key clinical questions.

DETAILED DESCRIPTION:
Lenvatinib was non-inferior to sorafenib in overall survival in untreated advanced hepatocellular carcinoma. The programmed cell death protein-1 (PD-1) antibody, was effective and tolerable in patients with hepatocellular carcinoma and portal vein tumor thrombus. We aimed to describe the efficacy and safety of Lenvatinib combined anti-PD1 antibody in patients with hepatocellular carcinoma who can not receive redical therapy.

ELIGIBILITY:
Inclusion Criteria:

1. HCC diagnosed by histopathological examination or Guidelines for Diagnosis and Treatment of Primary Liver Cancer or the recurrent HCC after surgery;
2. age between 18 and 75 years;
3. Stage B (middle stage) or C (late stage) HCC determined in accordance with Barcelona Clinic Liver Cancer staging system (BCLC stage). In case of stage B.
4. Previous use of any systemic therapy but intolerant, impotent or drug resistant.
5. Child-Pugh class A or B;
6. Eastern Cooperative Group performance status (ECOG) score of 0-2;
7. Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 32 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3
8. Prothrombin time ≤18s or international normalized ratio < 1.7.
9. Ability to understand the protocol and to agree to and sign a written informed consent document.

Exclusion Criteria:

1. Cholangiocellular carcinoma (ICC);
2. Patients with cancer thrombus in the main trunk of portal vein (Vp4), or cancer thrombus in inferior vena cava should be excluded;
3. The survival or patients less than 3 months.
4. Serious medical comorbidities.
5. Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
6. Known history of HIV
7. History of organ allograft
8. Known or suspected allergy to the investigational agents or any agent given in association with this trial.
9. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
10. Evidence of bleeding diathesis.
11. Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: For the advanced hepatocellular carcinoma (HCC), the targeted therapy and immunotherapy are recommended. This study focused on the management of Lenvatinib combined anti-PD1 antibody for the HCC. This study will create a database that will provide clinical parameters and outcomes of patients undergoing Lenvatinib and anti-PD1 antibody as part of their standard of care in hopes of answering key clinical questions.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Progression-Free-Survival(PFS) | 24 months
  Progression was defined as progressive disease by independent radiologic review according to mRECIST or death from any cause
Overall survival (OS) | 24 months
  OS is the length of time from the date of randomization until death from any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 6 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all randomized subjects whose best overall response (BOR) is either a CR or PR.
Disease control rate(DCR) | 24 months
  The proportion of patients who had a best response rating of complete response， partial response, or stable disease.
Adverse events | 24 months
  Safety will be evaluated according to the NCI CTCAE Version 4.03. All observations pertinent to the safety of the study medication will be recorded on the CRF and included in the final report.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No